CLINICAL TRIAL: NCT03953495
Title: BetterTogether: Evaluating the Health Effects of a Culturally Appropriate Web-based Relationship Education Tool That Targets Stigma-related Coping Behaviors in Rural Central Appalachian Female Same-Sex Couples
Brief Title: Better Together: A Web-based Relationship Education Tool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sharon Scales Rostosky (Other)
Responsible Party: Sponsor-Investigator, Sharon Scales Rostosky, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-0427-P4S
Record Dates: First submitted 2019-05-10; First posted 2019-05-16 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Same-Sex Relationships
Keywords: stress; stigma-related stress; relationship quality; depressive symptoms; anxiety; couples; intimate relationships; lesbian
MeSH Terms: conditions — Depression; Anxiety Disorders; Homosexuality, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Better Together (Experimental): Participants will be recruited with e-mail, print, and social media announcements and advertisements distributed through the professional contacts and networks of the investigators. The experimental group will consist of randomly assigned volunteers who meet the eligibility requirements (i.e., same-sex female couple over the age of 18 who lives in Central Appalachia).
  Interventions: Behavioral: Better Together

INTERVENTIONS:
Behavioral: Better Together — The Better Together Intervention consists of a 7 self-paced online relationship education modules. Following an introductory and overview module couples will complete each of the following together on their web-connected device (computer, ipad, phone). Each module includes didactic material, demonstration vignettes, and guided discussions or skills building exercises. Module 1 focuses on identifying individual and relationship strengths; Module 2 focuses on destructive communication patterns, Module 3 focuses on positive communication skills; Module 4 teaches a problem-solving technique; Module 5 focuses on stress and coping; Module 6 focuses on relationship expectations and commitment, and Module 7 provides a summary of the program. Each module takes approximately 30 minutes to an hour to complete. Metrics will be assessed at baseline, post-intervention, and at a 3 month follow up.

SUMMARY:
Health disparities have been documented in same-sex partnered women, including higher rates of cardiovascular disease, Type 2 diabetes, cancers, and mental health disorders. Higher rates of smoking, substance use, and obesity are behavioral risk factors that contribute to these chronic health problems. Living in rural areas with fewer social supports and less access to culturally sensitive healthcare services may also contribute to health disparities in sexual minorities. Their stigmatized identity is linked to minority stress, a well-documented social determinant of health behaviors and outcomes. Coping responses are an important couple-level mechanism that link stigma-related (minority) stress and health in same-sex couples. Relationship education (RE) programming is a potentially effective approach to increasing positive dyadic-level coping skills that support health. In a sample of 40 female same-sex couples, investigators will test the hypothesis that couples who complete newly revised, web-based RE modules that target health-related coping responses to stigma-related stress will report immediate (post-intervention) and persistent (3-month follow up) positive effects on their relationship quality (e.g., positive communication and problem-solving, relationship satisfaction, perceived partner support), stigma-related coping behaviors, and health (e.g., reduced substance use, depression/anxiety, physical health symptoms). This intervention represents one of the first efforts to test the effects of a culturally appropriate web-based relationship education tool that specifically targets health-related coping behaviors in rural female same-sex couples, a stigmatized, high-risk, under-researched and under-resourced population.

DETAILED DESCRIPTION:
Central Appalachian women in same-sex relationships experience health disparities. Higher rates of smoking, other substance use, and obesity are risk factors that contribute to health disparities in Central Appalachia women, and these health risk factors have been also been implicated in the health disparities faced by women who are same-sex partnered. In a national probability sample, lesbian and bisexual young adult women, compared to heterosexual young adult women, reported higher rates of smoking and heavy drinking, had significantly higher BMIs, and were significantly more likely to report an illness in the previous two weeks. The intervention in this pilot study is based on minority stress and relationship theories and current empirical findings reviewed below.

Stigma-related stress, a chronic form of social stress, largely accounts for health disparities.

Stigma affects health by creating conditions of chronic stress in those with stigmatized identities. This chronic (minority) stress has been linked to diminished mental and physical health. Specifically in rural LGB samples, stigma-related stress has been linked to higher levels of psychological distress (e.g., depression and anxiety), increased substance use, and overall poorer physical health, Same-sex couple members experience stigma-related stress because of experiences of discrimination and prejudice that targets them as individuals, as a couple, and, as a stigmatized social identity group. In their daily interactions, Central Appalachian same-sex couples experience discrimination and prejudice at work, in schools and churches, and in their families and communities. Even though same-sex couples in Central Appalachia can legally marry, stigma and discrimination persist. No state law in this region protects same-sex couples from discrimination in services, employment or housing.

The theory of minority stress as applied to LGB individuals describes a psychological process in which chronic experiences of prejudice and discrimination lead to fear and expectations of rejection, concerns about possible consequences of disclosing or concealing one's sexual minority identity or same-sex relationship, and internalized negativity or shame about one's relationship and one's identity. Minority stress among LGB-identified people appears to be on the increase nationally due to recent political events that threaten hard-won progress toward full equality of same-sex partnered individuals and their families.

Coping responses are an important mechanism that links stigma-related stress and health. To manage these chronic stigma-related stressors, LGB individuals use positive and/or negative coping responses that may buffer or exacerbate their effects of these stressors on health. Findings suggest that coping responses are an important mechanism linking stigma-related stress to poorer health outcomes. Therefore, helping this population to cope more effectively with stigma-related stress can buffer its negative health effects.

Same-sex couples share minority stress and strengths. Same-sex couples' relationships can simultaneously be the target of discrimination and prejudice and also the primary source of support for coping with that discrimination and prejudice. Conceptual models based in relationship science and minority stress theory and recent empirical evidence suggests that same-sex couples share minority stress. For example, when one couple member experiences discrimination at work, the minority stress that it triggers also affects the minority stress level of the other couple member. In other cases, the couple relationship itself is the target of discrimination, for instance, when extended family members refuse to accept the couple. Shared minority stress can take a toll on relationship quality unless couples find effective ways to cope. Distressed couples who rely on inadequate or unhealthy coping strategies are at risk for mental and physical health problems.

On the other hand, specific strengths and resiliencies enable same-sex couples to create satisfying and stable relationships even in the context of stigma-related stress. For example, female couples have demonstrated strengths in forming egalitarian partnerships that include sharing responsibility for the emotional climate of the relationship household and a commitment to supporting each other's health-related behaviors. Together these findings suggest the importance of intervening at the dyadic level by using couple-level strengths to enhance relationship skills and positive health-related coping behaviors to address stigma-related (minority) stress. Helping female same-sex couples to develop their relationship skills and use them to cope effectively with stigma-related stress in ways that support each other's health and well-being will help to address mental and physical health disparities in this population.

Relationship education (RE) programming is a potentially effective approach to increasing dyadic-level coping skills that support health-related behavior. Compared to different-sex couples, married/partnered sexual minority women receive less social support for their relationship from their families and communities, and as a result they tend to rely more heavily on their relationship for support. In addition to a lack of family and community support, same-sex couples in Central Appalachia often lack friendship networks that include other same-sex couples who could serve as role models and resources. Thus, Central Appalachia female same-sex couple can benefit from an accessible, evidence-based intervention that supports their relationship well-being, an important foundation for health.

In general, the purpose of RE is to increase knowledge and teach skills that will circumvent the development of severe problems in the future. RE programs have been shown to benefit married and unmarried different-sex couples across racial/ethnic and socio-economic backgrounds by effecting reliable change in communication and relationship satisfaction. Optimal RE programs should be tailored to the specific client population, accessible, grounded in theory and research, and directed at reducing risk factors and increasing protective factors at the individual and couple level. To date, RE programs have been limited to different-sex couples. Yet, prominent RE researchers have proposed the RE approaches that use same-sex couples' relationship skills and strengths to cope effectively with stigma-related stress are well-suited to support the health and well-being of these couples and their families. The current project builds upon and extends an RE workshop for female same-sex couples, which is based in relationship science and minority stress theory and has demonstrated post-intervention effects on relationship quality. In this randomized wait-list control trial, same-sex female couples achieved significant improvement in their relationship quality and communication skills that was maintained three months after the conclusion of the program. However, there was no evidence of program effects on stress or perceived support. Further, participants reported that the units on stress and social support were only somewhat helpful and could benefit from the inclusion of more specific strategies and skills. The current project will build upon and address limitations of previous research by piloting and testing the effectiveness of a revised program that uses newly developed modules to teach couples to use their relationship skills to cope with stigma-related stress in ways that support their long-term health and well-being (Aim 1).

Some evidence suggests that web-based relationship interventions (for different-sex couples) are superior to no treatment. In distressed different-sex couples, a web-based couple intervention significantly improved relationship quality and reduced pre-intervention symptoms of anxiety, depression, and physical health problems when compared to wait-list controls. The current project will extend previous work by adapting the revised RET to a web-based format to make it more accessible to rural female same-sex couples and evaluating feasibility, acceptability, adherence, and satisfaction (Aim 2).

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* self-identify as same-sex partnered
* female
* Central Appalachian resident

Exclusion Criteria:

* under 18 years old
* not currently in a committed relationship with a female partner
* identifies as male
* identifies as heterosexual
* has a male partner
* does not live in Central Appalachia
* does not have access to the internet and a computer or other device for completing the modules

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is investigating female same-sex relationships
Enrollment: 22 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2020-12-03 (Actual)

PRIMARY OUTCOMES:
Change in depression and anxiety. | up to 26 weeks
  Change in depression and anxiety will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) short form survey. Eight items measure depression symptom frequency over the past 7 days, and 8 items measure anxiety symptom frequency over the past 7 days. Each item is scored on a scale of 1 to 5 where 1 = never and 5 = always. A low cumulative score indicates low levels of anxiety/depression; a high cumulative score indicates high levels of anxiety/depression.
Health-related Quality of Life | up to 26 weeks
  This scale assesses the number of days out of 30 that the participant experienced poor physical health (0-30), poor mental health (0-30) and the number of days that poor physical or mental health kept them from working (0-30). Scores range from 0-90; lower scores indicating greater health-related quality of life.
Substance Use | up to 26 weeks
  Ten-item scale to assess substance use in the past 30 days. (Cigarette use/smoking: 3 items, Alcohol use (partner and self): 4 items, Marijuana use: 2 items, Prescription painkillers/opiates:1 item). Each item is scored on a frequency scale of 1-7, with 1 indicating less than once per month and 7 indicating more than once per day. Cumulative scores range from 10-70; higher scores indicate increased substance use.
Couples Satisfaction Index | up to 26 weeks
  Twelve-item scale assessing relationship satisfaction. Each item is scored on a scale of 1-7 where 1 = not at all satisfied and 7 = very satisfied. Average scores range from 1-7. An average score of 1 indicates low relationship satisfaction; an average score 7 indicates high relationship satisfaction.
Relationship Instability Index | up to 26 weeks
  Four-item scale assessing relationship instability. Each item is scored on a scale of 0 to 4 where 0 = Never; 1= Once or Twice; 2= Sometimes; 3= Often; 4 = Very Often. Cumulative scores range from 0-16. A cumulative score of 0 indicates low relationship instability; a cumulative score of 16 indicates high levels of relationship instability.
Relationship Confidence | up to 26 weeks
  Ten-item scale assessing relationship confidence. Each item is scored on a scale of 1 to 7 where 1 = Strongly Disagree and 7 = Strongly Agree. Average scores range from 1-7. An average score of 1 indicates low relationship confidence; an average score of 7 indicates high relationship confidence.
Couple Problem Solving | up to 26 weeks
  Six-item scale assessing couple problem solving. Each item is scored on a scale of 1 to 7 where 1 = Never Happens and 7 = Happens Most of the Time. Average scores range from 1-7. An average score of 1 indicates poor couple problem solving; an average score of 7 indicates good couple problem solving.
Couple Communication | up to 26 weeks
  Two combined subscales (27 items) measure the frequency of constructive and destructive conflict resolution behavior. Each item is scored on a scale of 1-7 where 1= Never Happens and 7 =Happens Most of the Time. Average scores range from 1-7. An average score of 1 indicates high levels of destructive conflict resolution behavior and low levels of constructive resolution behavior; an average score of 7 indicates low levels of destructive conflict resolution behaviors and high levels of constructive resolution behaviors.
Intimate Safety | up to 26 weeks
  Questionnaire (28-items) assessing intimate safety. Each item is scored on a scale of 0-4 where 0 = Never and 4 = Always. Average scores range from 0-4. An average score of 0 indicates low levels of intimate safety; an average score of 4 indicates high levels of intimate safety.
Relationship Dedication/Commitment | up to 26 weeks
  Eight-item scale assessing relationship dedication/commitment. Each item is scored on a scale of 1-7 where 1= Strongly Disagree and 7= Strongly Agree. Average scores range from 1-7. An average score of 1 indicates low levels of relationship dedication/commitment; an average score of 7 indicates high levels of relationship dedication/commitment.
Dyadic Coping | up to 26 weeks
  Fifteen-item scale measuring three types of dyadic coping: supportive coping by oneself (5 items), supportive coping of one's partner (5 items), and common dyadic coping (5 items). Each item is scored on a scale of 1-5 where 1= Very Rarely and 5= Very Often. Cumulative scores range from 15-75. A cumulative score of 15 indicates low levels of dyadic coping; a cumulative score of 75 indicates high levels of dyadic coping.
Perceived Relationship Marginalization | up to 26 weeks
  Four-item scale assessing perceived relationship marginalization. Each item is scored on a scale of 1-7 where 1= Very Much Disapproves and 7= Very Much Approves. Cumulative scores range from 4-28. A cumulative score of 4 indicates high levels of perceived relationship marginalization; a cumulative score of 28 indicates low levels of perceived relationship marginalization.
LGB Identity LGB Identity LGB Identity | up to 26 weeks
  Fifteen-item scale assessing feelings of positivity regarding lesbian, gay, or bisexual (LGB) identity. Each item is scored on a scale of 1-7 where 1= Strongly Disagree and 7 = Strongly Agree. Average scores range from 1-7. An average score of 1 indicates negative LGB identity; an average score of 7 indicates positive LGB identity.
Perceived Stress | up to 26 weeks
  Ten-item Cohen Perceived Stress Scale assessing the frequency of perceived stress over the past month. Each item is scored on a scale of 0-4 where 0= Never and 4= Very Often. Cumulative scores range from 0-40. A cumulative score of 0 indicates low perceived stress; a cumulative score of 40 indicates high perceived stress.
Coping Self-Efficacy | up to 26 weeks
  Thirteen-item scale assessing coping self-efficacy (6 problem solving items, 4 emotion-regulation items and 3 social support items). Each item is scored on a scale of 0-10 where 0= Cannot Do At All; 5= Moderately Certain Can Do; 10=Certain Can Do. Cumulative scores range from 0-130. A cumulative score of 0= low coping self-efficacy; a cumulative score of 130 indicates high coping self-efficacy.
Internalized Stigma (Public Identification) | up to 26 weeks
  Seven-item scale assessing public identification. Each item is measured on a scale of 1-7 where 1=Strongly Disagree and 7=Strongly Agree. Average scores range from 1-7. An average score of 1 indicates lower levels of internalized homophobia; an average score of 7 indicates higher levels of internalized homophobia.
Personal Feelings About Identity (Internalized Stigma) | up to 26 weeks
  Eight-item scale assessing public identification. Each item is measured on a scale of 1-7 where 1=Strongly Disagree and 7=Strongly Agree. Average scores range from 1-7. An average score of 1 indicates lower levels of internalized homophobia; an average score of 7 indicates higher levels of internalized homophobia
Mindful Self Care | up to 26 weeks
  Eighteen item scale assessing the frequency of self-care practices in the past 7 days using 3 subscales: physical care (8 items), mindful awareness (4 items) and mindful relaxation (6 items. Each item is scored on a scale of 0-4 where 0=Never (0 days); 1= rarely (1 day); 2= sometimes (2-3 days); 3= often (4-5 days); 4= regularly (6-7 days). On each subscale an average score of 0 indicates low frequency; an average score of 4 indicates high levels of self-care practice. A total score (sum of the subscale averages) of 0 indicates low levels of self-care practice; a score of 4 indicates high levels of self-care practice.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon S Rostosky, Ph.D., Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that underlie reported results published from this trial.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Three years after publication
Access Criteria: Access to data can be requested via email to PI.